CLINICAL TRIAL: NCT06660290
Title: A Phase 3b Study to Evaluate 0.003% AR-15512 Safety and Drop Attributes
Brief Title: A Study to Evaluate 0.003% AR-15512 Safety and Drop Attributes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEF512-E005
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye Disease
Keywords: Dry Eyes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Masking Description: In this single arm study, the subject is masked as to when they receive the Refresh Classic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- REFRESH® Classic, then 0.003% AR-15512 (Experimental): One drop of REFRESH® Classic ophthalmic solution administered topically to the eye, followed by 0.003% AR-15512 ophthalmic solution administered topically to the eye
  Interventions: Drug: 0.003% AR-15512 ophthalmic solution; Drug: REFRESH® Classic ophthalmic solution

INTERVENTIONS:
Drug: 0.003% AR-15512 ophthalmic solution — Investigational ophthalmic solution for topical instillation
Drug: REFRESH® Classic ophthalmic solution — Commercially available ophthalmic solution for topical instillation

SUMMARY:
The purpose of this study is to evaluate the proportion of ocular adverse events reported in subjects with dry eye disease (DED) between the intervention arm (0.003% AR-15512) and Refresh® Classic.

DETAILED DESCRIPTION:
This is a 1-visit study (Screening, Enrollment, Assessments).

ELIGIBILITY:
Key Inclusion Criteria:

* Corrected Visual Acuity (Snellen) 20/200 or better in both eyes;
* Good general and ocular health, as determined by the Investigator using medical history, ophthalmic examination and history;
* Capable of giving signed informed consent.

Key Exclusion Criteria:

* Current evidence of other clinically significant ophthalmic disease other than dry eye;
* History of ocular surgery within 1 year of the Study Visit;
* Use of any topical ocular anti-inflammatory medications (for example, Restasis®, Cequa™, Vevye™, Xiidra®), other prescription ophthalmic product for dry eyes, topical ocular corticosteroid, or non-steroidal-anti-inflammatory agents within 30 days of the Study Visit;
* Positive pregnancy test or currently breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Ocular Adverse Events | Day 1 post drop instillation
  Adverse Events are defined as any untoward medical occurrences associated with the administration of the study intervention in humans, whether or not considered to be related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (6):
- United States (6):
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Andover Eye Associates, Andover, Massachusetts
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No